CLINICAL TRIAL: NCT06581822
Title: Biomarkers for Pharmacoresponse in Bipolar Disorder - Coagulation
Status: Active, not recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Catharina Lavebratt Holmquist, Research group leader, Karolinska Institutet
Other Study IDs: 2023-04886-02
Record Dates: First submitted 2024-05-29; First posted 2024-09-03 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Previous studies indicate an association between severe psychiatric disorders, such as bipolar disorder, and increased risk of venous thromboembolism. However, to which extent this association is influenced by lithium treatment is currently unknown. In this prospective cohort study, the investigators aim to investigate the effect of bipolar disorder and lithium treatment on coagulation and the counterpart fibrinolysis.

DETAILED DESCRIPTION:
The investigators will analyse differences in coagulation

* using a case-control design where cases are bipolar patients not yet treated with lithium, and controls are healthy volunteers (Swedish ethical review authority Dnr 2023-05799-02, PI Kristoffer Månsson, KI).
* using a prospective cohort design, following the patients over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bipolar disorder but not yet treated with lithium, where there is a decision by the patient and the responsible doctor to start lithium treatment.

Exclusion Criteria:

* Inability to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bipolar disorder but not yet treated with lithium, where there is a decision by the patient and the responsible doctor to start lithium treatment. Patients are recruited in specialized care.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Extracellular vesicles | From enrollment to end of examination at 2 years
  Counts of plasma extracellular vesicles originating from blood platelets, leukocytes and vascular endothelial cells.
Hemostatic potential | From enrollment to end of examination at 2 years
  Overall hemostatic potential (OHP), coagulation potential (OCP) fibrinolytic potential (OFP) i citrate plasma.

OTHER OUTCOMES:
Plasma proteins of coagulation- or fibrinolysis-related processes | From enrollment to end of examination at 2 years
  Concentration in plasma of proteins involved in coagulation or fibrinolysis such as von Willebrand factor

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Not planning to share IPD